CLINICAL TRIAL: NCT02224872
Title: A Phase II Trial of Non-Myeloablative Conditioning and Transplantation of Partially HLA-Mismatched/Haploidentical Related or Matched Unrelated Bone Marrow for Patients With Refractory Severe Aplastic Anemia and Other Bone Marrow Failure Syndromes
Brief Title: Transplantation of Partially Mismatched Related or Matched Unrelated Bone Marrow for Patients With Refractory Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1424; IRB00031590 (Other: JHMIRB)
Record Dates: First submitted 2014-08-18; First posted 2014-08-25 (Estimated); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Severe Aplastic Anemia; Bone Marrow Failure Syndromes
Keywords: bone marrow transplant; thymoglobulin; cyclophosphamide; fludarabine; tacrolimus; Mycophenolic Acid Mofetil; chemotherapy; GVHD; haploidentical
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Failure Disorders | interventions — Bone Marrow Transplantation; thymoglobulin; fludarabine; Cyclophosphamide; Mesna; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone marrow transplant (Experimental): Thymoglobulin on days -9 to -7 Fludarabine on days -6 to -2 Cyclophosphamide on days -6, -5, 3, 4 TBI on day -1 BMT on day 0 Mesna on days 3, 4 Tacrolimus on days 5-365 Mycophenolic acid mofetil on days 5-35
  Interventions: Procedure: Bone marrow transplant; Drug: Thymoglobulin; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: TBI; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolic acid mofetil

INTERVENTIONS:
Procedure: Bone marrow transplant — Day 0
Drug: Thymoglobulin — 0.5 mg/kg IV on Day -9 2 mg/kg IV on Days -8, -7
Drug: Fludarabine — 30 mg/M2 IV on days -6 to -2
Drug: Cyclophosphamide — 14.5 mg/kg IV on days -6, -5, 3, 4
  Other Names: CTX
Radiation: TBI — 200 cGy on day -1
Drug: Mesna — 40 mg/kg IV on days 3, 4
Drug: Tacrolimus — For patients 18 years or older, tacrolimus will be given per institutional standards; may be increased or later changed to a PO BID schedule. Treatment to continue until Day 365 or longer if GVHD present
Drug: Mycophenolic acid mofetil — 15 mg/kg PO/IV TID beginning on day 5 through day 35
  Other Names: MMF

SUMMARY:
Our primary objective is to determine if it is feasible for SAA patients to be transplanted using non-myeloablative conditioning and post transplantation cyclophosphamide with partially HLA-mismatched donors.

DETAILED DESCRIPTION:
This research is being done to find out if bone marrow transplantation (BMT) followed by chemotherapy will help people with aplastic anemia who have failed other treatments.

You have a severe, life threatening disease (severe aplastic anemia) in your bone marrow. Your disease has come back or not responded after receiving one or more immunosuppressive treatments. High dose chemotherapy followed by bone marrow transplantation (BMT) has been used to treat blood diseases like yours but complications from Graft vs. Host disease (GVHD) and graft failure have limited the survival for those people.

A small study done at Johns Hopkins has shown that in subjects with other diseases (blood cancers) some immunosuppressive drugs given after the BMT have decreased how often subjects had complications of GVHD and engraftment failure.

People with aplastic anemia who have refractory disease (not responding to standard treatment) may join.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory SAA or very SAA defined:

  * Bone marrow (< 25% cellular)
  * Peripheral cytopenias (at least 2 of 3)

    * ANC < 500 per ml
    * Platelets < 20,000 per ml
    * Absolute retic < 60,000 or corrected retic < 1%
  * Very severe: as above, but ANC < 200
  * Disease may be designated as acquired or inherited if previous counts known (these other bone marrow failure disorders that are characterized by aplastic anemia may go by additional names such as dyskeratosis congenita or PNH)
  * Failed at least one course of immunosuppressive therapy (if presumed acquired disease). Patients with inherited disease will be characterized as refractory and do not require immunosuppressive first.
* Age 0- upper age limit as determined by current institutional standards
* Good performance status (ECOG 0 or 1; Karnofsky and Lansky 70-100)
* Patients and donors must be able to sign consent forms (or if a minor the parent will sign). Donors should be willing to donate.
* Patients must be geographically accessible and willing to participate in all stages of treatment.
* Adequate end-organ function as measured by:

  1. Left ventricular ejection fraction > or = to 35%, or shortening fraction > 25% (For pediatric patients, a normal ejection fraction is required)
  2. Bilirubin ≤ 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST ≤ 5 x ULN
  3. FEV1 and FVC > or = to 40% of predicted; or in pediatric patients, if unable to perform pulmonary function tests due to young age, oxygen saturation >92% on room air

Exclusion Criteria:

* Patients will not be excluded on the basis of sex, racial or ethnic background.
* Prior transfusions from selected donor (as this could have cause recipient alloimmunization against the donor)
* Women of childbearing potential who currently are pregnant (HCG+) or who are not practicing adequate contraception.
* Patients who have any debilitating medical or psychiatric illness that would preclude their giving informed consent or their receiving optimal treatment and follow up.
* Uncontrolled viral, bacterial, or fungal infections (HIV infection permitted if viral load undetectable)

Max Age: 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy DeZern, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] DeZern AE, Zahurak ML, Symons HJ, Cooke KR, Rosner GL, Gladstone DE, Huff CA, Swinnen LJ, Imus P, Borrello I, Wagner-Johnston N, Ambinder RF, Luznik L, Bolanos-Meade J, Fuchs EJ, Jones RJ, Brodsky RA. Haploidentical BMT for severe aplastic anemia with intensive GVHD prophylaxis including posttransplant cyclophosphamide. Blood Adv. 2020 Apr 28;4(8):1770-1779. doi: 10.1182/bloodadvances.2020001729. PMID 32343796

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone Marrow Transplant
Started | 18
Completed | 16
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 12
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 30 [5 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Is This Type of Transplantation for Severe Aplastic Anemia Feasible and Safe?
Description: Feasibility will be met with the following conditions: the patient has the transplant, is assessed for the safety endpoint, and survives one year. The safety monitoring plan is included to monitor graft failure (day 60), grade 2-4 acute graft versus host disease (day100), 6 month mortality (day 180), and chronic graft versus host disease (day 180).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 18

2. Secondary Outcome: Number of Patients That Have Survived at One Year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Number of Patients That Have Acheived Full Donor Chimerism by Day 60 After Transplant
Description: Donor chimerism will be measured in the peripheral blood around day 30 and day 60. Patients with >5% donor chimerism around day 60 will be considered as having engrafted.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 7

4. Secondary Outcome: Number of Patients That Expired Due to Non-relapsed-related Mortality Following Transplant
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 0

5. Secondary Outcome: Number of Participants With Major Toxicities Related to Transplant
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 0

6. Secondary Outcome: Number of Patients That Expired Due to Transplant Related Mortality
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 0

7. Secondary Outcome: Number of Patients With Primary or Secondary Graft Failure Following Transplant
Description: Graft failure: < 5% donor chimerism in blood and/or bone marrow on ~Day 30 or after and on all subsequent measurements.
  Primary graft failure: < 5% donor chimerism in blood and/or bone marrow by ~ Day 56 Secondary graft failure: achievement of > 5% donor chimerism, followed by sustained <5% donor chimerism in blood and/or bone marrow.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 17

8. Secondary Outcome: Number of Participants With Grade II-IV or Grade III-IV Acute GVHD
Description: Participants were graded during clinical visits based on evidence and extent of skin rash, liver involvement, and GI tract involvement
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 17

9. Secondary Outcome: Participants With Chronic GVHD at One Year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 3

10. Secondary Outcome: Length of Time Required for Patients to Recover ANC and Platelet Counts After Transplant
Description: CBC drawn daily with a WBC differential once the total WBC is greater than 100 until ANC > 500 for three days or two consecutive measurements over a three day period; then CBC drawn weekly with differential.
Time Frame: 1 year
Measure: Median (Full Range); unit: days
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
days | 18.85 [14 to 48]

11. Secondary Outcome: Participants That Were GVHD Free, Relapse Free Survival (GRFS)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 18
Participants | 14

ADVERSE EVENTS:
Time Frame: Adverse event data will be collected from day 0 of transplant through day 60 post transplant. All-Cause mortality is reported up to one year after transplant
Arm/Group | Bone Marrow Transplant
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Transplant (N=18)
Acute Respiratory Distress Syndrom (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intracranial Hemorrhage (Vascular disorders) | 1 (1)
Retroperitoneal Hemorrhage (Vascular disorders) | 1 (1)
Hemorrhagic Shock (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Persistent Fevers (Infections and infestations) | 1 (1)
dysuria/hematuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT02224872/Prot_SAP_000.pdf